CLINICAL TRIAL: NCT02212353
Title: Care Delivery in Acute Hospital Settings: an Observational Study. WP1 P3
Brief Title: Care Delivery in Acute Hospital Settings: an Observational Study
Acronym: PERFECTED
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: DTC-RP-PG-0311-12004
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Dementia; Hip Fractures
MeSH Terms: conditions — Dementia; Hip Fractures | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Site 1 Health Care Professionals: Observational research. This is a cohort of health care professionals working in site 1 in delivering to care to neck of femur patients.
  Interventions: Other: Observational study, not interventional
- Site 2 Health Care Professionals: Observational research. This is a cohort of health care professionals working in site 2 in delivering to care to neck of femur patients.
  Interventions: Other: Observational study, not interventional
- Site 3 Health Care Professionals: Observational research. This is a cohort of health care professionals working in site 3 in delivering to care to neck of femur patients.
  Interventions: Other: Observational study, not interventional

INTERVENTIONS:
Other: Observational study, not interventional

SUMMARY:
This small observational study is a contractual component of a 5-year (2013-18) NIHR funded programme called PERFECTED (Peri-operative Enhanced Recovery hip FracturE Care of paTiEnts with Dementia) whose overall aim is to develop and pilot an evidence-based intervention to improve the hospital care of patients with dementia suffering a fractured hip. The findings from this particular observational study will support other PERFECTED work-packages in establishing current care practices in acute hospital settings for older people in general with hip fractures.

Observation is a well-established qualitative technique widely used to understand cultures, processes and interactions in defined locations including hospitals. In this study, researchers will observe day-to-day practices on specific ortho-geriatric wards and Emergency Departments in three English hospitals (Norfolk and Norwich University Hospital, Bradford Royal Infirmary and Queen's Medical Centre in Nottingham). Observations will occur intermittently over a 4-week period, covering the full 24h cycle. The prime objective of the study is to describe delivery of care to older patients with a hip fracture including an assessment of cost consequences. Crucially, the observations will focus exclusively upon the hospital personnel that routinely provide care in the designated locations being observed. Other individuals who frequent the locations (patients, visitors and other more peripheral health care professionals) are NOT the focus of the research and will be regarded as "incidental others" rather than "participants". This approach is common in observational research.

Observations will be conducted by experienced qualitative researchers and assisted by specifically trained lay researchers to provide a valuable service-user dimension to the study. Field-notes and contextual information will be collected and thematically analysed, again in partnership with trained 'lay' researchers. Resulting data will address the pre-defined aims of the observational study and feed into the findings reported across the whole of work package 1 of PERFECTED.

DETAILED DESCRIPTION:
Rationale and background information

Hip fracture

Hip fracture is a common orthopaedic injury amongst older adults. It is estimated that more than 1.2 million individuals will suffer hip fracture annually worldwide (Gullberg et al, 1997) and this total is expected to surpass 6 million by the year 2050 (Cooper et al, 1992; Odén et al, 2013). Hip fracture has a significant impact on the health and independence of patients and their families, with an increased risk of functional decline, admission to long-term care institutions and high mortality rates within the first 12 months post-fracture (Seitz et al, 2011). Furthermore the economic implications for the NHS are significant in both direct and indirect costs (Hernlund et al, 2013).

People with dementia

It is estimated that 25% of all beds in UK acute hospital wards are occupied by people with dementia (PwD) (Royal College of Psychiatrists 2009). Improving acute hospital care for PwD is high on the national agenda, as this group is particularly vulnerable to poor quality care and adverse outcomes (NHS Confederation 2010). Patients with dementia - primarily older people, are highly susceptible to insensitive care as complex needs in relation to their memory, thinking, orientation, comprehension, calculation, learning capability, language, and judgment are often unrecognised and unaddressed (Alzheimer Society 2009). Older people and their families consistently place high value on hospital care which promotes personalised relationships between patients and staff. This is particularly pertinent for people with impaired cognition or communication difficulties ( Alzheimer Society 2009).

People with hip fracture and dementia

People with dementia (PwD) have a four-fold increased risk of a hip fracture compared to matched cognitively intact cohorts (Gruneir et al, 2010; Laditka et al, 2005). Identifying the needs of people with dementia can be difficult. Engagement and progress with post-operative hip fracture rehabilitation can also be compromised for patients with dementia. Data suggests that clinical outcomes (incidence of delirium, mortality and post-operative complication rates) are poorer for PwD following hip fracture when compared to cognitively intact individuals (Smith et al, 2013).

Enhanced Recovery Pathways

The process of "Enhanced Recovery" was developed in Denmark by Prof Kehlet and has been used in the UK since the early 2000s (Department of Health 2013a). It is an integrated, multi-modal, evidence-based approach that enables hospital patients to recover from surgery, treatment or illness more effectively and leave hospital sooner. Since their formal introduction into the NHS in 2009, Enhanced Recovery Pathways (ERP) are becoming standard practice for many elective surgical operations and have resulted in a reduction in both length of hospital stays and readmission rates while generating high levels of patient satisfaction (Department of Health 2013a).

Enhanced Recovery Pathways (ERP) for elective surgery are becoming more common and there is an increasing commitment to drive the delivery of enhanced recovery as standard practice (Department of Health 2013a). ERP in acute hip fracture is much rarer. The pathways are typically structured around six discrete phases which follows the patients' journal from hospital arrival through to discharge, these are:

* Emergency Department - arrival and diagnoses
* Pre-operative - ward admittance and preparation for operation
* Intra-operative - the operation
* Post-operative - recovery from the operation
* Rehabilitation - optimising recovery of function
* Discharge - return to home or appropriate residence

These pathways are based upon evidence-based, documented national and internationally expert guidelines and are subject to frequent clinical review. A key co-morbidity that is recognised is cognitive impairment and as described above clinical outcomes for PwD can be significantly worse to non-cognitively impaired patients. Following National Guidelines on Dementia Care (Department of Health 2009a) most acute hospital Trusts are implementing general dementia care strategies throughout hospitals. Given that the proportion of patients dementia that sustain hip fractures is increasing year on year, some experts (McGilton et al 2013) have suggested that the subgroup of patients with dementia and hip fracture should have a specific treatment pathway, to acknowledge the clear differences in presentation and care needs. Developing an ERP specifically for patients with dementia and hip-fracture is the precise objective of the overall PERFECTED research programme.

The PERFECTED research programme

The PERFECTED (Peri-operative Enhanced Recovery hip FracturE Care of paTiEnts with Dementia) research programme was awarded to Dr Chris Fox (UEA) in November 2013. This is a 5 year project funded under the National Institute for Health Research (NIHR) Programme Grant for Applied Research initiative. For a summary of the accepted research proposal please see annex 1. The overall aim of PERFECTED is to improve hospital care for PwD admitted with a fractured hip. The research will first develop and then examine the feasibility, acceptability and potential clinical and cost effectiveness of an optimised "enhanced recovery pathway" (ERP) for these patients. The PERFECTED programme is structured as 4 Work Packages (WPs); the primary aims of each are as follows:

* WP1: to establish best practice and define an ERP for patients with hip fracture and dementia in acute hospitals.
* WP2: to determine the staff training and cultural/organisational changes required to implement and maximise adherence to the aforementioned ERP.
* WP3: to undertake a pilot study to assess the clinical and cost effectiveness of the ERP that will inform the design of a future definitive Randomised Controlled Trial.
* WP4: to disseminate the data and lessons learned from the programme and develop a definitive trial proposal.

This protocol relates to phase 3 of WP1 only. This specific phase is an observational study and involves researchers observing care delivery in specified ortho-geriatric wards at the Norfolk and Norwich University Hospital (NNUH), the Queen's Medical Centre (QMC) Nottingham and the Bradford Royal Infirmary (BRI). Observations will also take place in the Emergency Department (ED) of each of these hospitals on an opportunistic basis. Observations will occur in each of the sites intermittently over a 4-week period sequentially and will cover the full 24h cycle. That is, we will do 4 weeks of observations at the NNUH, before moving to BRI and observing for 4 weeks, and then finish by undertaking 4 weeks of observations at QMC. Data elicited from these observations will address this study's research aims and will also inform the wider aims of WP1 by describing the context (including cost consequences) of care delivery to hospital patients with hip fracture, some of whom will have dementia. It is essential to emphasise that although PERFECTED overall (including WP1) is concerned with older hip-fracture patients who have dementia, phase 3 WP1 (this observational study) is concerned with all older hip-fracture patients in general.

As a research programme PERFECTED is iterative. To create one total ethical protocol would not be feasible. We will be submitting numerous protocols in line with the programme's development. The aims, procedures and ethical considerations associated with phase 3 WP1, the observational study, are the sole objectives of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Health Care Professioanls delivering care in the observational environments

Exclusion Criteria:

* Those who are not Health Care Professioanls delivering care in the observational environments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Secondry Care
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2014-12-12 (Actual); Study Completion 2014-12-16 (Actual)

PRIMARY OUTCOMES:
To observe and describe the general day-to-day practices and routines in three English acute hospitals for treating older patients with hip fracture. | Observations in each of the 3 sites will take place for a 4 week period.
  The overall aim of this study (phase 3, WP1 of PERFECTED) is to observe and describe the general day-to-day practices and routines in three English acute hospitals for treating older patients with hip fracture. The influence on care practices of significant co-morbidities, particularly dementia, will especially be noted. Observations will take place in defined areas on specified ortho-geriatric wards and in EDs. The study's aims and objectives focus on the delivery of care. As such, the focus of the observations is solely upon those health professionals who routinely deliver care in the designated spaces.

CONTACTS AND LOCATIONS:
Overall Officials: George C Fox, Principal Investigator — University of East Anglia